CLINICAL TRIAL: NCT02406963
Title: Photographic Email Correspondence for Pediatric Urology Post-Operative Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster Children's Hospital (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Mandy Rickard, Nurse Practitioner, McMaster Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-169
Record Dates: First submitted 2015-03-23; First posted 2015-04-02 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Post-Operative Complication; Pediatric Urology
Keywords: telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TTC (Active Comparator): Current standard of care- a telephone call with the NP in the event of a post-operative concern where advice/interventions/reassurance is provided based on information provided by family
  Interventions: Other: Telephone Call
- PEC (Experimental): Experimental arm, the standard telephone call with the NP and the addition of a digital photograph of the surgical site for assessment prior to the administration of advice
  Interventions: Other: Digital Photograph; Other: Telephone Call

INTERVENTIONS:
Other: Digital Photograph — A digital photograph sent by the family of the surgical site
  Arms: PEC
Other: Telephone Call — Standard telephone call with the nurse practitioner

SUMMARY:
A pilot research study is planned to occur within the pediatric urology service the spring of 2015. All pediatric urology patients in the immediate post-operative period of 0-14 days will be eligible for this study. This study will compare the current standard of care for managing post-operative complications (a telephone conversation with the NP) versus an experimental intervention (telephone call and an electronic photograph of the surgical site). Before the surgical patient is discharged from the hospital, consent will be obtained for participation. Once a family initiates contact with the NP with a post-operative concern they will be randomized to either the control or the experimental group. Those in the control group will receive the current standard of care, which is telephone advice only. Those in the experimental group will speak to the NP on the telephone and will be requested to send an electronic photograph of their child's surgical site to the NP for assessment and advice. Photographs will be assessed using a standardized tool by both NPs and this information will be entered into a database. The investigators will be measuring the number of emergency department (ED) and/or unplanned clinic visits in both groups. An unplanned clinic visit is defined as a visit that is required due to an unexpected complication or concern before the original scheduled post-operative follow-up as determined by the surgeon. The investigators will be tracking the number of follow-up phone calls for both groups, as well as requiring participants to complete a family/patient experience survey after speaking to the NP.

DETAILED DESCRIPTION:
This study design will be a pilot randomized controlled trial. Consent for this study will be obtained within the circle of care immediately before the patient is discharged home following surgery. The families will be instructed to contact the NP by telephone with any post-operative questions or concerns they have about their child. Once the family initiates contact with the NP, they will be randomized into either the experimental (PEC) group or the control (TTC) group.

Once randomization has occurred, the NP will obtain all necessary information from the parent by addressing all points in expertise based script developed by the Pediatric Urology Team for both groups. Those randomized to the control group (TTC) will be provided recommendations based on information obtained during the standard telephone call. Families who are randomized into the PEC (experimental) group will be required to send a digital photograph of the child's surgical site to the professional email address of NP. Should they agree to send digital photographs they will be required to give consent for email correspondence, which will be emailed to them by the NP. Once they have consented they may send digital photographs to the NP of their child's surgical site, which will be assessed by both NPs using an expertise-based assessment tool. This information will be entered into REDCap. The NPs will come to a unanimous decision regarding advice to be provided and this will be communicated to the parents. Upon completion of the interaction with the NP the RA will contact the family to complete the family/patient experience survey over the telephone. Family/patient experience will be measured using an adapted validated tool "Nurse Practitioner Satisfaction Survey" consisting of 10 questions directly related to telephone interaction with the NP. This survey consists of a Likert Scale with scores ranging from 1-5 with 5 being the most positive response. Follow up telephone calls for both groups will be logged in MediTech as well as the RedCAP database. All telephone calls will be documented within the MediTech system and included in patient's chart in order to maintain current standard of care. All digital photos will be printed and placed in the patient's chart and deleted from the email server, which is the current process for those engaging in PEC.

Recruitment for this study will occur for 7 months with the aim of recruiting 40 patients per arm in order to obtain the feasibility data. However, a sample size calculation has been carried out and assuming 75% power and an alpha error of 5% using a one sided test, the required sample size to answer the definitive research question is 114 patients per group.

Data will be analyzed by comparing the number of ED and unplanned clinic visits for both groups, as well as the number of follow up phone calls received. This will be done using descriptive statistics and a t-test for independent means. Family/patient experience will also be measured between the two groups (PEC and TTC) using descriptive statistics and a t-test for independent means. Subgroup analysis will be done to determine which subgroup of post-operative patients benefit most from PEC (i.e., penile surgeries).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-17 years who have undergone urological surgery.
* Children within the immediate post-operative period (0-14 days).
* Children with concerns directly related to operative site including, but not limited to catheters, stents, rashes and urine output.

Exclusion Criteria:

* Surgical patients outside the immediate post-operative period.
* Those families who are unwilling or unable to email digital photographs.
* Concerns related to issues other than the operative site (medications, follow up appointments, return to activities).
* Inability to understand written consent due to language barrier

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Feasibility Data- Recruitment Rate | 7 Months
  Recruitment rate over 7 month enrollment period to help determine whether recruitment for a larger scale trial will be feasible
Feasibility Data- Survey Completion | One Year
  Participants compliance with completing the patient experience questionnaire after discussion with the NP.
Feasibility Data- Engagement rate of participants in sending photos via email | One Year
  Measuring the compliance and willingness of participants to send digital photos of surgical site to NP in order to determine if larger scale trial is feasible

SECONDARY OUTCOMES:
Number of ED/ unplanned clinic visits in the PEC group compared to those in TTC group | One Year
Number of follow up phone calls received from each group | One Year
Comparing family experience of both groups | One Year
  Families will complete validated questionnaire after speaking to the NP on teh phone to evaluate experience. Both groups will complete this questionnaire and responses compared.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Rickard, MN-NP, Principal Investigator — McMaster Children's Hospital
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada